CLINICAL TRIAL: NCT01855204
Title: Low Tube Voltage Computed Tomographic (CT) Urography Using Low Concentration Iodine Contrast Agent: a Comparison Study With Conventional CT Urography
Brief Title: Low Tube Voltage Computed Tomographic (CT) Urography Using Low Concentration Iodine Contrast Agent
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Yeon Cho, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: SeoulNUH-rad
Record Dates: First submitted 2013-04-27; First posted 2013-05-16 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Exposure to Medical Diagnostic Radiation
Keywords: Computed Tomography, Spiral; Urography; Radiation dosage; Contrast media

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional (Active Comparator): Computed tomographic urography was done with conventional protocols.
  Interventions: Radiation: Computed tomographic urography
- Reduced (Experimental): Computed tomographic urography was done with the protocols of low voltage and low iodine concentration.
  Interventions: Radiation: Computed tomographic urography

INTERVENTIONS:
Radiation: Computed tomographic urography — Computed tomographic (CT) urography was done with the protocols of low voltage and low iodine concentration.

SUMMARY:
Computed Tomographic (CT) urography is the best imaging modality to evaluate obstructing lesions of urinary tract such as urinary stone, tumor and inflammatory lesion. The purpose of our study is to compare images of CT urography performed by low voltage and low concentrated iodine CT contrast with them of conventional CT urography.

DETAILED DESCRIPTION:
Computed Tomographic (CT) urography is the best imaging modality to evaluate obstructing lesions of urinary tract such as urinary stone, tumor and inflammatory lesion. It is needed that CT urography should have the high contrast between target lesion described as filling defect and adjacent contrast filled urinary tract. For the implementation of high contras, conventional CT urography has been performed with higher voltage and higher concentrated CT contrast than another CT protocols. The higher voltage results in the more radiation exposure. And the intravenous injection of higher concentrated CT contrast results in the increase of the prevalence of contrast induced nephrotoxicity.

The purpose of our study is to compare images of CT urography performed by low voltage and low concentrated iodine CT contrast with them of conventional CT urography.

ELIGIBILITY:
Inclusion Criteria:

* Patients to perform Computed Tomographic (CT) urography
* Patients without diminish of renal function (serum creatinine: more than 1.4 mg/dl & glomerular filtration rate: more than 34 mL/min/1.73 m2)

Exclusion Criteria:

* patients to have operations and/or injuries of urinary system
* patients to have the histories of anaphylaxis or allergic reaction about intravenous iodine contrast material

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-02 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Measurement of Radiation Dose | The day of admission (within 24hours)

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Yeon Cho, Professor, Principal Investigator — Departement of Radiology, Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea